CLINICAL TRIAL: NCT00718991
Title: A Physician Initiated Prospective Multicenter Study on Excimer Laser Recanalisation in the Treatment of Long Infrapopliteal Lesions in Patients With Critical Limb Ischemia
Brief Title: EXCimEr Laser for Long lENgTh Lesions in Below-The-Knee Arteries Study
Acronym: EXCELLENT-BTK
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: too slow enrollment
Sponsor: Flanders Medical Research Program (Network)
Collaborators: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-005
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: CLI; excimer laser; debulking
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): CLI patients receiving excimer laser recanalisation for the treatment of long infrapopliteal lesions
  Interventions: Device: Spectranetics Turbo elite™ excimer laser catheter

INTERVENTIONS:
Device: Spectranetics Turbo elite™ excimer laser catheter — The Spectranetics Turbo elite™ excimer laser catheters are percutaneous intravascular devices constructed of multiple optical fibers around a guidewire lumen. The laser catheters transmit ultraviolet energy from the Spectranetics CVX-300® Excimer Laser System to the obstruction in the artery. The ultraviolet energy is delivered to the tip of the laser catheter to photo-ablate fibrous, calcific and atheromatous lesions, thus recanalizing diseased vessels.

SUMMARY:
This investigation is designed to assess the immediate and long-term angiographic patency outcomes of excimer laser recanalisation followed by PTA in the treatment of long (>50 mm) infrapopliteal lesions in patients with critical limb ischemia (CLI)

The Spectranetics Turbo elite™ excimer laser catheters are percutaneous intravascular devices constructed of multiple optical fibers around a guidewire lumen. The laser catheters transmit ultraviolet energy from the Spectranetics CVX-300® Excimer Laser System to the obstruction in the artery. The ultraviolet energy is delivered to the tip of the laser catheter to photo-ablate fibrous, calcific and atheromatous lesions, thus recanalizing diseased vessels.

ELIGIBILITY:
Inclusion Criteria:

* The treatment vessel is DeNovo
* Stenotic (>50%) or occlusive atherosclerotic disease of infrapopliteal artery(s)
* Length of target lesion is > 50 mm
* Reference target vessel diameter between 2-4.0 mm by visual assessment
* Documented Rutherford Class 4 or 5 symptomatic critical limb ischemia
* The patient must be >18 years of age
* Life-expectancy of more than 12 months
* The patient has no child bearing potential or negative serum pregnancy test within 7 days of the index procedure
* The patient must be willing and able to return to the appropriate follow-up times for the duration of the study
* The patient must provide written patient informed consent that is approved by the ethics committee
* Anatomic Inclusion Criteria

  * All inflow lesions successfully (<30 residual stenosis) treated prior to target lesion treatment during same procedure or according standard of care without unresolved complications
  * At least one angiographically visible target at the ankle for establishment of straight line flow.

Exclusion Criteria:

* Patient refusing treatment
* The target vessel segment diameter is not suitable for available catheter design.
* Unsuccessfully treated endovascular or bypass( >30% residual stenosis) proximal ( iliac, SFA, popliteal) inflow limiting arterial/graft stenosis
* Lesion lies within or adjacent to an aneurysm
* The patient has a known allergy to heparin, Aspirin or other antiaggregant therapies or a bleeding diatheses or is unable, or unwilling, to tolerate such therapies.
* The patient has a history of prior life-threatening contrast media reaction.
* The patient is currently enrolled in another investigational device or drug trial.
* The patient is currently breast-feeding, pregnant or intends to become pregnant.
* The patient is unable to provide informed consent
* The patient has end stage renal disease (currently on any form of dialysis)
* Known Left Ventricular Ejection Fraction < 35%
* The patient has had an MI within 30 days prior to enrollment
* The patient has had a CVA within 90 days prior to enrollment
* Serum Creatinine > 150 µmol
* The patient has a previous bypass in the target limb
* The patient has a current systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Angiographic patency for laser + PTA, as defined by < 50% stenosis in the target lesion with straight line flow to the foot | 12 months
Absence of Major Adverse Events defined as death, amputation of treated limb and target vessel revascularization | 6 months

SECONDARY OUTCOMES:
Immediate angiographic laser recanalization success + PTA, defined as a residual diameter stenosis ≤30% and absence of flow-limiting dissection on visual assessment after combined excimer laser and PTA recanalization treatment | Procedure
Absence of Major Adverse Events defined as death, amputation of treated limb and target vessel revascularization | 12 months
Limb-salvage rate at all follow-up visits, defined as lack of major amputation of treated limb. Limb-salvage rate (LSR) is defined as 1 minus major amputation rate | 12 months
Serious adverse events defined as being fatal, life-threatening, or judged to be severe by the investigator; result in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged or new hospitalization | 12 months
Clinical success at follow-up is defined as an improvement of Rutherford classification of one class or more as compared to the pre-procedure Rutherford classification | 12 months
Health Economics assessment being: length of hospital stay, duration of the procedure, unplanned visits, retreatment and diagnostic procedure codes, material and medication costs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Peeters, MD, Principal Investigator — Imelda Hospital, Bonheiden, Belgium; Marc Bosiers, MD, Principal Investigator — AZ St-Blasius, Dendermonde, Belgium
Locations (2):
- Belgium (2):
  - Imelda Hospital, Bonheiden
  - AZ St-Blasius, Dendermonde